CLINICAL TRIAL: NCT00843466
Title: Compatibility of a Mild, Moisturizing Hand Cleanser for Patients With Mild to Moderate Hand Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00002004; 31963
Record Dates: First submitted 2008-06-02; First posted 2009-02-13 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Hand Dermatosis
Keywords: Hand dermatitis
MeSH Terms: conditions — Hand Dermatoses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild moisturizing Hand Cleanser (Active Comparator): The test group will be provided with a mild moisturizing hand cleanser for all hand cleansing needs during the duration of the study.
  Interventions: Other: Mild, moisturizing hand cleanser
- Current Hand Cleanser (No Intervention): The control group will continue to use their current cleanser for all hand washing.

INTERVENTIONS:
Other: Mild, moisturizing hand cleanser — Hand cleanser ingredient list:
  Ammonium Lauryl Sulfate, Ammonium Laureth Sulfate, Cocamide MEA, PEG-5 Cocamide Cocamidopropyl Betaine Sodium Lauroyl Sarcosinate Glycerin Petrolatum Soybean Oil Sodium Hydroxypropyl Starch Phosphate Lauric Acid Lauryl Alcohol PEG-14M Guar hydroxypropyl trimonium chloride DMDM Hydantoin; Iodopropynyl Butylcarbamate Etidronic Acid Tetrasodium EDTA Titanium Dioxide Fragrance Sodium Hydroxide Water
  Arms: Mild moisturizing Hand Cleanser

SUMMARY:
The purpose of this study is to find out if the use of a hand cleanser that adds moisture to the skin will help improve skin rashes caused by frequent hand washing (hand dermatitis).

DETAILED DESCRIPTION:
The objective of this protocol is to evaluate compatibility and potential benefits of daily use of a marketed mild, moisturizing hand cleanser for subjects/patients who experience mild to moderate hand dermatitis induced by frequent cleansing.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* In general good health
* Hands free of cuts and abrasions
* Agree to adhere to the requirements listed in the informed consent
* Willing and able to use a mild, moisturizing, non-antibacterial cleanser for all hand washing purposes for the duration of the test period
* Willing to refrain from participating in any other clinical research trial for the duration of the study

Exclusion Criteria:

* Documented allergies to study product components, soaps, latex, or fragrances
* History of the following conditions which may affect the response of the skin or the interpretation of the results: insulin dependent diabetes, or peripheral vascular diseases
* Participating in a concurrent clinical study involving treatment of your hands
* Currently using a prescription medication for hand dermatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from May 22,2007 to May 12, 2008 at Wake Forest University in Winston Salem.
Groups:
- Test Product: The test group was provided with a test product for all hand cleansing needs during the duration of the study.
- Control Group (Current Product): The control group continued to use their current cleanser for hand washing.
Period: Overall Study
Arm/Group | Test Product | Control Group (Current Product)
Started | 24 | 18
Completed | 24 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Control Group (Current Product) | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 18 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 45 [18 to 78] | 40 [20 to 65] | 41 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 24 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment
Description: Changes in global disease severity on a scale from 0-4 with 0 being clear and 4 being severe
Time Frame: Wk 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mild Moisturizing Hand Cleanser Test Product: The test group was provided with a test product for all hand cleansing needs during the duration of the study.
- No Treatment: The control group continued to use their current cleanser for hand washing.
Arm/Group | Mild Moisturizing Hand Cleanser Test Product | No Treatment
Number analyzed (Participants) | 24 | 18
units on a scale | 1.0 [0.8 to 1.2] | 1.1 [0.7 to 1.4]

ADVERSE EVENTS:
Arm/Group | Test Product | Control Group (Current Product)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 0/24 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No